CLINICAL TRIAL: NCT02105233
Title: Brain Mimicking Fluid. Improving Ultrasound Images in Brain Tumor Surgery With the Use of Brain Mimicking Fluid: a Preliminary Technical and Safety Study
Brief Title: Improving Ultrasound Images in Brain Tumor Surgery With the Use of Brain Mimicking Fluid
Acronym: BMF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: National Competence Services for Ultrasound and Image-guided Therapy (Unknown); SINTEF Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/1266; 2012-005567-27 (EudraCT Number)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Brain Neoplasms; Glioma
Keywords: ultrasonography; ultrasonics; brain; surgery
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMG (Experimental): brain mimicking fluid
  Interventions: Biological: brain mimicking fluid

INTERVENTIONS:
Biological: brain mimicking fluid — filled into the operation cavity during surgery for glioblastoma
  Other Names: acoustic fluid

SUMMARY:
Prognosis in patients with glioblastomas (the most aggressive high-grade glioma) remains unfavourable. Tools for improving brain tumor surgery, in particular for gliomas, are increasing. There seems to be an agreement that achieving extensive resections, when done safely without jeopardizing neurological function, improves survival.

Ultrasound is currently used as a tool for providing 2D or 3D images for the purpose of tumor localization and resection control. For the use in resection control the resection cavity is filled with saline to provide acoustic coupling between the ultrasound transducer and tissue. However, attenuation of acoustic waves is very low in saline compared to the brain and this difference in attenuation is the cause of artifacts that may severely degrade the ultrasound images. Such artifacts are seen as high-intensity signal at the resection cavity wall and beyond, potentially masking small tumor remnants and generally making the interpretation of images more difficult.

This research group has developed an acoustic fluid intended for use in the resection cavity instead of saline. Tests in laboratory measurements have shown that the fluid reduces artifacts and has the potential to enhance ultrasound image quality in brain tumor surgery. The investigators expect that the acoustic fluid will make it easier to detect small tumor remnants near the end of an operation, thus increasing success of glioma surgery. The purpose of this study is to test the fluid during surgery for histopathologically proven glioblastoma to assess safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* A glioblastoma is suspected when there is a solitary brain tumour with ring-like contrast enhancement and oedema with no recent history (last 3 years) of primary tumour elsewhere
* In cases where histopathology is not known from previous biopsy or resection (i.e. diagnosis is suspected based on MRI findings and not from previous surgery) a tissue sample for frozen section is necessary. The fluid will only be used in cases where glioblastoma is suggested from this preliminary histopathological assessment.

Exclusion Criteria:

* Intended biopsy only (meaning: cases not suitable for resection)
* Other entities than glioblastoma is suspected
* Allergy to diary products and marine products
* Hypersensitvity to egg protein
* Hypersensitivity to soya or peanut protein
* Hypersensitvity to glycerol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
adverse events | 1-72 hours
  All adverse events registered but with special emphasis on:
  Intraoperatively -- epileptic seizures Immidiate postoperative -- hydrocephalus (MR images), imflammation of tissue that was in contact with AF (MR images)
adverse events | 1 month
  All adverse events registered but with special emphasis on:
  hydrocephalus (MR images) inflammation (MR images)
adverse events | 6 months
  All adverse events registered but with special emphasis on:
  hydrocephalus (MR images), inflammation (MR images)
adverse events | up to 6 months
  All adverse events registered but with special emphasis on:
  unusual clinical events, neurological deterioration or reduced consciousness

SECONDARY OUTCOMES:
image quality | 1 day
  during the operation
  * Qualitative score of ultrasound image quality (poor-medium-good)
  * Qualitative score of artefacts in ultrasound images (none-some-much)
image signal-to-noise ratio | 1 day
  after the operation: image analysis by quantitative measurements of signal-to-noise ratio (SNR)

CONTACTS AND LOCATIONS:
Overall Officials: Geir Bråthen, phd md, Study Director — St. Olavs Hospital
Locations (1):
- Department of Neurosurgery, St Olavs Hospital, Trondheim, Norway